CLINICAL TRIAL: NCT05911308
Title: A Pilot Window of Opportunity Study Evaluating Durvalumab (MEDI4736) in Combination With Platinum Doublet Chemotherapy Followed by Evaluation of Durvalumab (MEDI4736) in Combination With Platinum Doublet Chemotherapy and Abequolixron (RGX-104) in Non-small Cell Lung Cancer
Brief Title: Abequolixron (RGX-104) and Durvalumab in Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor is closing the trial.
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: AstraZeneca (Industry); Rgenix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2113
Record Dates: First submitted 2023-06-09; First posted 2023-06-22 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Neoadjuvant therapy; abequolixron (RGX-104); LXR/ApoE; carboplatin; abraxane; pemetrexed
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; Carboplatin; SB 742881; Albumin-Bound Paclitaxel; Taxes; 130-nm albumin-bound paclitaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant therapy (Experimental): Subjects with operable Non-Small Cell Lung Cancer received neoadjuvant durvalumab plus platinum doublet chemotherapy and neoadjuvant durvalumab plus platinum doublet chemotherapy in combination with abequolixron (RGX-104), an LXR/ApoE agonist.
  Interventions: Drug: Durvalumab; Drug: Carboplatin; Drug: Abequolixron; Drug: Abraxane; Drug: Pemetrexed

INTERVENTIONS:
Drug: Durvalumab — 1,500 mg Durvalumab IV infusion will be given on day 1 of each cycle for 3 cycles.
  Other Names: Imfinzi
Drug: Carboplatin — Carboplatin IV infusion will be given on day 1 of each cycle for 3 cycles. The dose will be AUC 5.
  Other Names: Paraplatin
Drug: Abequolixron — 100 or 120 mg Abequolixron will be administered by mouth twice a day for 5 days followed by 2 days off throughout your treatment (5 days a week for up to 9 weeks).
  Other Names: RGX 104; RGX-104; RGX104; SB-742881
Drug: Abraxane — 100 mg/m2 Abraxane will be given by IV infusion on days 1, 8, and 15 of each cycle for 3 cycles.
  Other Names: Paclitaxel albumin-bound; Nab-paclitaxel
Drug: Pemetrexed — 500 mg/m2 pemetrexed will be given by IV infusion on day 1 of each cycle for 3 cycles.
  Other Names: Alimta

SUMMARY:
Non-Small Cell Lung Cancer (NSCLC) is one of the deadliest types of cancer. In lung cancer patients with a tumor that can be removed by surgery, adjuvant chemotherapy increases survival. Neoadjuvant therapy may have advantages such as, it may be more tolerable prior to surgery, earlier treatment may be more efficacious, and it can provide an indication of treatment response. Neoadjuvant treatment can provide pre- and post-treatment specimens for correlative analysis to better understand mechanisms of action and resistance.

This pilot study will investigate the effects of neoadjuvant durvalumab plus platinum doublet chemotherapy and neoadjuvant durvalumab plus platinum doublet chemotherapy in combination with abequolixron (RGX-104), an LXR/ApoE agonist, in subjects with NSCLC who are scheduled to undergo surgical resection as part of their standard of care.

The purpose of this study is to study how well using a combination of durvalumab, platinum doublet chemotherapy (carboplatin/abraxane or carboplatin/pemetrexed), and abequolixron treats non-small cell lung cancer before surgery. Durvalumab (a type of immunotherapy) and platinum doublet chemotherapy are drugs that are individually approved for use during the treatment of cancer. FDA (Food and Drug Administration) has not approved the combined use of these drugs in treating non-small cell lung cancer. Abequolixron is not FDA approved for the treatment of cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent obtained to participate in the study and

   HIPAA authorization for the release of personal health information.
2. Age ≥ 18 years at the time of consent.
3. Histologically or cytologically confirmed non-small cell lung cancer for which surgical resection

   would be standard of care.
4. ECOG Performance Status of 0-1
5. Body weight of > 40 kg
6. Is able to swallow and retain oral medication.

Exclusion Criteria:

1. Participation in another clinical study with an investigational product during the last 3 weeks
2. Concurrent enrollment in another clinical study unless it is an observational (non-interventional)

   clinical study or during the follow-up period of an interventional study.
3. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment with the

   exception of those mentioned in this protocol. Concurrent use of hormonal therapy for noncancer-

   related conditions (e.g., hormone replacement therapy) is acceptable.
4. Lack of full recovery from a major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP.
5. History of allogenic organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Feasibility of surgery | Up to 120 days
  Feasibility will be evaluated as the delay time between the completion of neoadjuvant therapy and surgery. A failure of feasibility will be defined as a delay in the planned surgery of more than 42 days (surgical delay of 35 days, plus 7 days for scheduling).

SECONDARY OUTCOMES:
Toxicities | Up to 1 years after surgery
  Toxicities related to study treatment therapy will be classified and graded according to The NCI Common Terminology Criteria for Adverse Events (NCI-CTCAE v5.0).
  NCI-CTCAE v5.0 is a descriptive terminology that can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Major pathologic response rate - squamous histology | Up to 120 days
  Major pathologic complete response rate after neoadjuvant chemotherapy will be assessed via surgical pathology report in subjects with non-small cell lung carcinoma - squamous histology.
  Major pathologic response is defined as equal to or less than 10% residual tumor following neoadjuvant therapy.
Major pathologic response rate - non squamous histology | Up to 120 days
  Major pathologic complete response rate after neoadjuvant chemotherapy will be assessed via surgical pathology report in subjects with non-small cell lung carcinoma - nonsquamous histology.
  Major pathologic response is defined as equal to or less than 10% residual tumor following neoadjuvant therapy.
Pathologic complete response rate (PCR) -durvalumab in combination with platinum doublet chemotherapy | Up to 120 days
  PCR -durvalumab in combination with platinum doublet chemotherapy will be histologically evaluated at the time of surgery, in subjects receiving neoadjuvant treatment with durvalumab in combination with platinum doublet chemotherapy.
  Pathologic complete response (pCR) is the disappearance of all signs of cancer in tissue samples removed during surgery or biopsy (pT0). Also called pathologic complete remission. Pathologic Partial Response (pPR), is the presence of only non-invasive cancer in tissue samples (<pT2)
Pathologic complete response rate (PCR) - durvalumab in combination with platinum doublet chemotherapy plus abequolixron | Up to 120 days
  Pathologic complete response rate (PCR) - durvalumab in combination with platinum doublet chemotherapy plus abequolixron will be histologically evaluated at the time of surgery, in subjects receiving neoadjuvant treatment with durvalumab in combination with platinum doublet chemotherapy plus abequolixron.
  Pathologic complete response (pCR) is the disappearance of all signs of cancer in tissue samples removed during surgery or biopsy (pT0). Also called pathologic complete remission. Pathologic Partial Response (pPR), is the presence of only non-invasive cancer in tissue samples (<pT2)
Clinical response rate (CRR) - durvalumab in combination with platinum doublet chemotherapy | Up to 1 years after surgery
  CRR is defined as the clinical response rate is the combination of complete response (CR) + partial response (PR) defined by The overall response rate will be assessed per Response Evaluation Criteria Solid Tumors (RECIST) 1.1 in subjects receiving durvalumab in combination with platinum doublet chemotherapy.
  Based on RECIST v1.1, Complete Response (CR) is the Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; and Overall Response Rate (ORR) = CR + PR/total number of subjects.
Clinical response rate (CRR) - durvalumab in combination with platinum doublet chemotherapy plus abequolixron | Up to 1 years after surgery
  CRR is defined as the clinical response rate is the combination of complete response (CR) + partial response (PR) defined by The overall response rate will be assessed per Response Evaluation Criteria Solid Tumors (RECIST) 1.1 in subjects receiving durvalumab in combination with platinum doublet chemotherapy plus abequolixron.
  Based on RECIST v1.1, Complete Response (CR) is the Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; and Overall Response Rate (ORR) = CR + PR/total number of subjects.
Recurrence-free survival (RFS) - durvalumab in combination with platinum doublet chemotherapy | Up to 5 years
  RFS - durvalumab in combination with platinum doublet chemotherapy will be defined as the time from the time after surgery to disease recurrence or death (whichever occurs first) and will be defined by RECIST 1.1. in subjects receiving neoadjuvant therapy with durvalumab in combination with platinum doublet chemotherapy.
  Based on RECIST v1.1 Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), no response or less response than Partial or Progressive; or Progressive Disease (PD), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Recurrence-free survival (RFS)- durvalumab in combination with platinum doublet chemotherapy plus abequolixron | Up to 5 years
  RFS - durvalumab in combination with platinum doublet chemotherapy will be defined as the time from the time after surgery to disease recurrence or death (whichever occurs first) and will be defined by RECIST 1.1. in subjects receiving neoadjuvant therapy with durvalumab in combination with platinum doublet chemotherapy plus abequolixron
  Based on RECIST v1.1 Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), no response or less response than Partial or Progressive; or Progressive Disease (PD), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Overall Survival (OS) - durvalumab | Up to 5 years
  OS - durvalumab is defined as the time from the first day of study therapy to the date of death for any cause, in subjects receiving neoadjuvant therapy with durvalumab in combination with platinum doublet chemotherapy.
Overall Survival (OS) - durvalumab in combination with platinum doublet chemotherapy plus abequolixron | Up to 5 years
  OS - durvalumab in combination with platinum doublet chemotherapy plus abequolixron is defined as the time from the first day of study therapy to date of death for any cause, in subjects receiving neoadjuvant therapy with durvalumab in combination with platinum doublet chemotherapy plus abequolixron.

CONTACTS AND LOCATIONS:
Overall Officials: Jared Weiss, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials